CLINICAL TRIAL: NCT01519570
Title: Use of an Electronic Medical Record to Improve Standard Practice in the Primary Care Setting: A Randomized-Controlled Study of Herpes Zoster Vaccination Rates
Brief Title: Use of an Electronic Medical Record in the Primary Care Setting to Improve Herpes Zoster Vaccination Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Stuart Beatty, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010H0290
Record Dates: First submitted 2012-01-12; First posted 2012-01-27 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2018-08

CONDITIONS: Herpes Zoster Disease
Keywords: Herpes Zoster vaccine; Electronic patient portal; Electronic medical record; Primary care; Immunizations
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- An informational packet regarding shingles and the HZV (Experimental)
  Interventions: Other: An informational packet regarding shingles and the HZV was sent to patients identified by the EMR
- Standard medical care from their primary care physician (No Intervention)

INTERVENTIONS:
Other: An informational packet regarding shingles and the HZV was sent to patients identified by the EMR — The EMR generated a list of patients aged 60 or older without HZV documentation. Patients were categorized into two subgroups based on activated electronic patient portal (EPP) status. Randomized patients from each subgroup received an informational packet regarding shingles and the HZV by either the EMR or USPS mail, depending on EPP status. A pharmacist reviewed the medical chart of interested patients to assess if the HZV was clinically indicated; eligible patients were mailed a HZV prescription.
  Arms: An informational packet regarding shingles and the HZV

SUMMARY:
Despite the significant benefits of herpes zoster vaccine (HZV), vaccination rates remain low. Electronic medical records (EMR) can serve as a practical strategy to better facilitate the application of preventative health care, such as increasing immunization rates. A new care model that can increase the herpes zoster vaccination rate, as well as other preventative health services, is warranted. The objective of this study is to investigate if the functions of an EMR, in combination with a pharmacist as part of the care team, can improve the herpes zoster vaccination rate.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 60 years of age

Exclusion Criteria:

* Documented herpes zoster vaccine in the EMR

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2589 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Beatty, PharmD, Principal Investigator — Ohio State University; Shelley H Otsuka, PharmD, Study Chair — The Ohio State Univeristy; Neeraj H Tayal, MD, Study Chair — Ohio State University; Kyle Porter, MAS, Study Chair — Ohio State University; Peter J Embi, MD, MS, Study Chair — Ohio State University
Locations (1):
- The Ohio State University Martha Morehouse General Internal Medicine Clinic, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | An Informational Packet Regarding Shingles and the HZV | Standard Medical Care From Their Primary Care Physician
Started | 500 | 2089
Completed | 500 | 2089
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | An Informational Packet Regarding Shingles and the HZV | Standard Medical Care From Their Primary Care Physician | Total
Number analyzed (Participants) | 500 | 2089 | 2589
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 500 | 2089 | 2589
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (9.4) | 73.1 (8.1) | 72.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 265 | 1174 | 1439
  Male | 235 | 915 | 1150
Region of Enrollment [Number; unit: participants]
  United States | 500 | 2089 | 2589

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received the Herpes Zoster Vaccine
Description: Six months after the intervention, a second EMR report was generated to determine the change in vaccination rate of both the intervention and control groups.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | An Informational Packet Regarding Shingles and the HZV | Standard Medical Care From Their Primary Care Physician
Number analyzed (Participants) | 500 | 2089
Participants | 500 | 2089

2. Secondary Outcome: Difference in Vaccination Rates Between Patients Who Recieved a Mailed Letter Versus a Secure Email
Description: Difference in vaccination rates between patients sent communications via US postal service (USPS) and those sent communications via electronic patient portal (EPP)
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Amount of Time Required by a Clinical Pharmacist to Manage This Workflow
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | An Informational Packet Regarding Shingles and the HZV | Standard Medical Care From Their Primary Care Physician
Serious Adverse Events (participants affected / at risk) | 0/500 | 0/2089
Other Adverse Events (participants affected / at risk) | 0/500 | 0/2089

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes